CLINICAL TRIAL: NCT03844321
Title: Healthy Mind Healthy You: A Study of Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of South Florida (Other); Global Healthy Living Foundation (Other); University of North Carolina (Other); University of California, Los Angeles (Other); Genetic Alliance (Other); COPD Foundation (Other); The Duchenne Registry (Other); University of California, San Francisco (Other); Children's Hospital Medical Center, Cincinnati (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Accelerated Cure Project for Multiple Sclerosis (Other); Mayo Clinic (Other); Phelan-McDermid Syndrome Foundation (Other); Immune Deficiency Foundation (Other); Brigham and Women's Hospital (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Dauten Family Center for Bipolar Treatment Innovation, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001648
Record Dates: First submitted 2017-10-31; First posted 2019-02-18 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Stress
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): 8 sessions of online mindfulness-based cognitive therapy
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Brief Mindfulness (Experimental): 3 sessions of online mindfulness therapy
  Interventions: Behavioral: Brief Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — 8 sessions of online mindfulness-based cognitive therapy
  Arms: Mindfulness-Based Cognitive Therapy
Behavioral: Brief Mindfulness — 3 sessions of online mindfulness therapy
  Arms: Brief Mindfulness

SUMMARY:
Most people experience stress at some point in their lives. Stress, especially when severe, can not only make you feel bad, it can also worsen existing health problems like heart disease, type 2 diabetes, obesity, high blood pressure, depression, and even cancer. Healthy Mind, Healthy You is a new study about how mindfulness can help people cope with stress. Funded by the Patient Centered Outcome Research Institute (PCORI) and involving 19 Patient Powered Research Networks (PPRNs), Healthy Mind Healthy You will be able to study the effects of mindfulness on a wide variety of populations and conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must be a member (patient/member of special population or caregiver) of one of the 19 PCORI Patient-Powered Research Networks (PPRN)
* Must be age 18 or older

Exclusion Criteria:

* Under the age of 18 years
* Unable to read, understand, and/or participate in mindfulness exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4412 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Nierenberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sylvia LG, Lunn MR, Obedin-Maliver J, McBurney RN, Nowell WB, Nosheny RL, Mularski RA, Long MD, Merkel PA, Pletcher MJ, Tovey RE, Scalchunes C, Sutphen R, Martin AS, Horn EJ, O'Boyle M, Pitch L, Seid M, Redline S, Greenebaum S, George N, French NJ, Faria CM, Puvanich N, Rabideau DJ, Selvaggi CA, Yu C, Faraone SV, Venkatachalam S, McCall D, Terry SF, Deckersbach T, Nierenberg AA. Web-Based Mindfulness-Based Interventions for Well-being: Randomized Comparative Effectiveness Trial. J Med Internet Res. 2022 Sep 12;24(9):e35620. doi: 10.2196/35620. PMID 36094813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals from 17 Patient Centered Outcomes Research Institute (PCORI) Patient Powered Research Networks (PPRNs) who were over the age of 18, able to read and understand English, and/or participate in mindfulness exercises were eligible to participate in Healthy Mind Healthy You Study. Participants were recruited through each PPRN. Recruitment for the study occurred from 2/27/2019 to 10/1/2019 and the follow up period ended on 1/31/2020.
Pre-assignment Details: This study was inclusive of all subgroups, with the exception of individuals under the age of 18 or and individuals not able to participate in mindfulness exercises, with broad inclusion and minimal exclusion criteria. Participants' date of birth which was checked for accuracy by the data management system. After consent, participants completed baseline questionnaires on their mindfulness practices in the past, stress, anxiety, well-being, psychosocial functioning and PPRN-specific assessments.
Period: Overall Study
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Started | 2220 | 2192
Completed | 579 | 533
Not Completed | 1641 | 1659

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness | Total
Number analyzed (Participants) | 2220 | 2192 | 4412
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.95 (14.72) | 54.63 (15.05) | 55.29 (14.90)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex Assigned at Birth
  Participants
    Female | 1780 | 1768 | 3548
    Male | 429 | 410 | 839
    Other | 0 | 1 | 1
    Ambiguous | 6 | 5 | 11
    Unknown | 5 | 8 | 13
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender Identity
  Participants
    Woman | 1690 | 1654 | 3344
    Man | 402 | 388 | 790
    No selected answer | 49 | 43 | 92
    Genderqueer | 32 | 39 | 71
    Transgender male/Trans man/Female-to-male | 17 | 32 | 49
    Prefer not to answer | 6 | 10 | 16
    Other | 8 | 8 | 16
    Something else | 4 | 8 | 12
    Multiple gender categories | 5 | 4 | 9
    Transgender female/Trans woman/Male-to-female | 6 | 4 | 10
    Unknown | 1 | 2 | 3
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sexual Orientation
  Participants
    Straight | 1816 | 1744 | 3560
    Bisexual | 91 | 102 | 193
    Gay | 72 | 78 | 150
    Lesbian | 69 | 78 | 147
    Queer | 56 | 67 | 123
    No selected answer | 39 | 35 | 74
    Prefer not to answer | 24 | 30 | 54
    Asexual | 18 | 22 | 40
    Multiple sexual orientations | 14 | 8 | 22
    Something else | 5 | 14 | 19
    Questioning | 9 | 7 | 16
    Other | 3 | 6 | 9
    Unknown | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Origin
  Participants
    White | 1957 | 1917 | 3874
    Multiple Race | 68 | 59 | 127
    Black, African American, African, or AfroCaribbean | 45 | 52 | 97
    Asian | 39 | 38 | 77
    No selected answer | 36 | 41 | 77
    Prefer not to answer | 24 | 43 | 67
    Other | 32 | 24 | 56
    Native American, American Indian, or Alaska Native | 12 | 15 | 27
    Unknown | 5 | 2 | 7
    Native Hawaiian or other Pacific Islander | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Non-Hispanic | 2078 | 2042 | 4120
    Hispanic | 101 | 97 | 198
    No selected answer | 20 | 22 | 42
    Prefer not to answer | 16 | 24 | 40
    Other | 2 | 5 | 7
    Unknown | 3 | 2 | 5
World Health Organization-5 Well-Being Index [Mean (Standard Deviation); unit: units on a scale] — This 5-item questionnaire assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being.
  units on a scale | 50.2 (20.6) | 50.6 (20.7) | 50.4 (20.7)
Five Facet Mindfulness Questionnaire [Mean (Standard Deviation); unit: units on a scale] — This 39-item questionnaire examines five aspects of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Only the questions related to non-judging of inner experience and non-reactivity were administered (15 items total). The total score on these 15 items was used (range: 15-75). Higher scores represent greater mindfulness.
  units on a scale | 49.9 (11.2) | 49.9 (11.0) | 49.9 (11.1)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — This 10-item questionnaire evaluates an individual's experiences of stress in the previous month. Scores range 0-40, with higher scores representing greater perceived stress.
  units on a scale | 20.1 (3.71) | 20.2 (3.64) | 20.2 (3.67)
PROMIS Emotional Distress - Anxiety Short Form (Adult, 4-Item) [Mean (Standard Deviation); unit: units on a scale] — This 4-item questionnaire measures self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal in the past seven days. Scores range 4-20, with higher scores representing more severe anxiety symptoms.
  units on a scale | 8.94 (3.64) | 8.98 (3.61) | 8.96 (3.62)
PROMIS Emotional Distress - Depression Short Form (Adult, v. 8a) [Mean (Standard Deviation); unit: units on a scale] — This 8-item questionnaire measured perceived depressive symptoms over the past week. Scores range 8-40, with higher scores representing more severe depressive symptoms.
  units on a scale | 16.4 (7.00) | 16.3 (7.07) | 16.4 (7.04)
PROMIS: Ability to Participate in Social Roles and Activities Short Form (Adult, 4-item) [Mean (Standard Deviation); unit: units on a scale] — This 4-item questionnaire measures the perceived ability to perform one's everyday social roles and activities. Scores range 4-20 with higher scores representing fewer limitations (greater abilities).
  units on a scale | 10.6 (4.35) | 10.6 (4.29) | 10.6 (4.32)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Weekly Change on World Health Organization-5 (WHO-5)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. We used linear mixed effects models to examine the effect of the interventions on weekly WHO-5 scores. Change = estimated average weekly change during time frame.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in scale score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in scale score
  Baseline to 8 Weeks | 0.78 [0.63 to 0.93] | 0.76 [0.60 to 0.91]
  Baseline to 20 Weeks | 0.41 [0.34 to 0.48] | 0.33 [0.26 to 0.40]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; We used a linear mixed effects model to examine the difference in effect of time on weekly WHO-5 scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 8 weeks. This model accounts for the covariance of repeated measurements within subjects, and we used maximum likelihood estimation to adjust for missing assessment scores. The model includes a random slope and intercept, and fixed effects for intervention, time, and an intervention by time interaction; Test type: Superiority; p = .820, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; df = 1607; Difference in Slopes = -0.02, 95% CI 2-sided [-0.24 to 0.19] — Slope estimate = difference in slopes between conditions (Mindfulness Light vs. Mindfulness-Based Cognitive Therapy) during time frame
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; We used a linear mixed effects model to examine the difference in effect of time on weekly WHO-5 scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 20 weeks. This model accounts for the covariance of repeated measurements within subjects, and we used maximum likelihood estimation to adjust for missing assessment scores. The model includes a random slope and intercept, and fixed effects for intervention, time, and an intervention by time interaction; Test type: Superiority; p = .110, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1147; Difference in Slopes = -0.08, 95% CI 2-sided [-0.18 to 0.02] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Estimated Weekly Change on Perceived Stress Scale (PSS)
Description: The PSS is a 10-item questionnaire that evaluates an individual's experiences of stress in the previous month. Scores range 0-40, with higher scores representing greater perceived stress. Change = estimated average weekly change during time frame.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in scale score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in scale score
  Baseline to 8 Weeks | -0.13 [-0.16 to -0.09] | -0.15 [-0.18 to -0.12]
  Baseline to 20 Weeks | -0.08 [-0.09 to -0.06] | -0.07 [-0.08 to -0.05]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PSS scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 8 weeks; Test type: Superiority; p = .284, Mixed Models Analysis — A two-sided significance level of .05 was used; df= 1726; Difference in Slopes = -0.03, 95% CI 2-sided [-0.07 to 0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PSS scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 20 weeks; Test type: Superiority; p = .394, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1018; Difference in Slopes = 0.01, 95% CI 2-sided [-0.01 to 0.03] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Estimated Weekly Change on Patient Reported Outcomes Measurement Information System (PROMIS): Emotional Distress-Depression Short Form
Description: The PROMIS: Emotional Distress-Depression Short Form is an 8-item questionnaire that measures perceived depressive symptoms over the past week. Scores range 8-40, with higher scores representing more severe depressive symptoms. Change = estimated average weekly change during time frame.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in scale score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in scale score
  Baseline to Week 8 | -0.19 [-0.23 to -0.15] | -0.17 [-0.21 to -0.12]
  Baseline to Week 20 | -0.11 [-0.13 to -0.09] | -0.06 [-0.08 to -0.04]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PROMIS: Emotional Distress-Depression Short Form scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 8 weeks; Test type: Superiority; p = .431, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1591; Difference in Slopes = 0.03, 95% CI 2-sided [-0.04 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PROMIS: Emotional Distress-Depression Short Form scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 20 weeks; Test type: Superiority; p < .001, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1159; Difference in Slopes = 0.05, 95% CI 2-sided [0.02 to 0.08] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Estimated Weekly Change on Patient Reported Outcomes Measurement Information System (PROMIS): Emotional Distress-Anxiety Short Form
Description: The PROMIS: Emotional Distress-Anxiety Short Form is a 4-item questionnaire that measures self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal in the past seven days. Scores range 4-20, with higher scores representing more severe anxiety symptoms. Change = estimated average weekly change during time frame.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in scale score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in scale score
  Baseline to Week 8 | -0.12 [-0.15 to -0.10] | -0.13 [-0.16 to -0.11]
  Baseline to Week 20 | -0.07 [-0.08 to -0.06] | -0.05 [-0.06 to -0.04]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PROMIS: Emotional Distress-Anxiety Short Form scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 8 weeks; Test type: Superiority; p = .399, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1601; Difference in Slopes = -0.01, 95% CI 2-sided [-0.05 to 0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PROMIS: Emotional Distress-Anxiety Short Form scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 20 weeks; Test type: Superiority; p = .048, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1171; Difference in Slopes = 0.02, 95% CI 2-sided [0.00 to 0.03] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Estimated Weekly Change on Patient Reported Outcomes Measurement Information System (PROMIS): Ability to Participate in Social Roles and Activities Short Form
Description: The PROMIS: Ability to Participate in Social Roles and Activities Short Form is a 4-item questionnaire that measures the perceived ability to perform one's everyday social roles and activities. Scores range 4-20 with higher scores representing fewer limitations (greater abilities). Change = estimated average weekly change during time frame.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in scale score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in scale score
  Baseline to Week 8 | -0.12 [-0.15 to -0.09] | -0.14 [-0.17 to -0.11]
  Baseline to Week 20 | -0.05 [-0.06 to -0.04] | -0.04 [-0.06 to -0.03]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PROMIS: Ability to Participate in Social Roles and Activities Short Form scores (reverse scored) in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 8 weeks; Test type: Superiority; p = .488, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1560; Difference in Slopes = -0.02, 95% CI 2-sided [-0.06 to 0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly PROMIS: Ability to Participate in Social Roles and Activities Short Form scores (reverse scored) in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 20 weeks; Test type: Superiority; p = .446, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1179; Difference in Slopes = 0.01, 95% CI 2-sided [-0.01 to 0.03] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Estimated Weekly Change on Five Facet Mindfulness Questionnaire (FFMQ) Abbreviated
Description: The FFMQ is a 39-item questionnaire that examines five aspects of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Only the questions related to non-judging of inner experience and non-reactivity were administered (15 items total). The total score on these 15 items was used (range: 15-75). Higher scores represent greater mindfulness. Change = estimated average weekly change during time frame.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in scale score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in scale score
  Baseline to 8 Weeks | 0.92 [0.84 to 1.00] | 0.88 [0.79 to 0.96]
  Baseline to 20 Weeks | 0.43 [0.39 to 0.46] | 0.37 [0.34 to 0.41]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used a linear mixed effects model to examine the difference in effect of time on weekly FFMQ scores in Mindfulness Light vs. Mindfulness-Based Cognitive Therapy conditions from baseline to 8 weeks; Test type: Superiority; p = .469, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1618; Difference in Slopes = -0.04, 95% CI 2-sided [-0.16 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; As with the primary outcome, we used linear mixed effects models to examine the effect of time on weekly FFMQ scores across both intervention conditions from baseline to 20 weeks; Test type: Superiority; p = .033, Mixed Models Analysis — A two-sided significance level of .05 was used; df = 1067; Difference in Slopes = -0.06, 95% CI 2-sided [-0.11 to -0.01] — [estimate comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Age
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Age was self-reported.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: Age 45 | 0.98 [0.78 to 1.19] | 0.75 [0.55 to 0.95]
  Baseline to 8 Weeks: Age 55 | 0.81 [0.66 to 0.96] | 0.73 [0.58 to 0.89]
  Baseline to 8 Weeks: Age 65 | 0.64 [0.48 to 0.80] | 0.72 [0.54 to 0.90]
  Baseline to 20 Weeks: Age 45 | 0.53 [0.43 to 0.63] | 0.38 [0.29 to 0.48]
  Baseline to 20 Weeks: Age 55 | 0.44 [0.36 to 0.51] | 0.33 [0.25 to 0.40]
  Baseline to 20 Weeks: Age 65 | 0.34 [0.27 to 0.42] | 0.27 [0.19 to 0.35]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Age measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .046, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Age measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .275, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

8. Other Pre Specified Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Baseline Perceived Stress Scale (PSS)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. The PSS is a 10-item questionnaire that evaluates an individual's experiences of stress in the previous month. Scores range 0-40, with higher scores representing greater perceived stress.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Median (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to Week 8: PSS = 18 | 0.64 [0.48 to 0.80] | 0.61 [0.44 to 0.78]
  Baseline to Week 8: PSS = 20 | 0.78 [0.63 to 0.93] | 0.75 [0.60 to 0.90]
  Baseline to Week 8: PSS = 22 | 0.92 [0.75 to 1.09] | 0.89 [0.71 to 1.07]
  Baseline to Week 20: PSS = 18 | 0.35 [0.27 to 0.42] | 0.28 [0.21 to 0.36]
  Baseline to Week 20: PSS = 20 | 0.42 [0.35 to 0.48] | 0.33 [0.25 to 0.40]
  Baseline to Week 20: PSS = 22 | 0.48 [0.40 to 0.57] | 0.37 [0.28 to 0.45]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PSS measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .977, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PSS measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .341, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

9. Other Pre Specified Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Baseline Patient Reported Outcomes Measurement Information System (PROMIS): Emotional Distress-Depression Short Form (PROMIS: EDD)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. The PROMIS: EDD is a 4-item questionnaire that measures self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal in the past seven days. Scores range 4-20, with higher scores representing more severe anxiety symptoms.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to Week 8: PROMIS: EDD = 10 | 0.51 [0.32 to 0.70] | 0.47 [0.28 to 0.66]
  Baseline to Week 8: PROMIS: EDD = 15 | 0.72 [0.57 to 0.86] | 0.69 [0.54 to 0.84]
  Baseline to Week 8: PROMIS: EDD = 20 | 0.92 [0.75 to 1.10] | 0.91 [0.73 to 1.09]
  Baseline to Week 20: PROMIS: EDD = 10 | 0.30 [0.21 to 0.39] | 0.26 [0.17 to 0.34]
  Baseline to Week 20: PROMIS: EDD = 15 | 0.39 [0.32 to 0.46] | 0.31 [0.23 to 0.38]
  Baseline to Week 20: PROMIS: EDD = 20 | 0.48 [0.39 to 0.56] | 0.36 [0.27 to 0.44]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PROMIS: EDD measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .885, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PROMIS: EDD measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .319, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

10. Other Pre Specified Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Baseline Patient Reported Outcomes Measurement Information System (PROMIS): Emotional Distress-Anxiety Short Form (PROMIS: EDA)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. The PROMIS: EDA is a 4-item questionnaire that measures self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal in the past seven days. Scores range 4-20, with higher scores representing more severe anxiety symptoms.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: PROMIS: EDA = 5 | 0.46 [0.26 to 0.66] | 0.47 [0.26 to 0.68]
  Baseline to 8 Weeks: PROMIS: EDA = 10 | 0.85 [0.68 to 1.01] | 0.83 [0.66 to 0.99]
  Baseline to 8 Weeks: PROMIS: EDA = 15 | 1.23 [0.91 to 1.55] | 1.18 [0.86 to 1.50]
  Baseline to 20 Weeks: PROMIS: EDA = 5 | 0.25 [0.16 to 0.35] | 0.18 [0.08 to 0.28]
  Baseline to 20 Weeks: PROMIS: EDA = 10 | 0.46 [0.38 to 0.53] | 0.37 [0.29 to 0.45]
  Baseline to 20 Weeks: PROMIS: EDA = 15 | 0.66 [0.50 to 0.81] | 0.56 [0.40 to 0.72]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PROMIS: EDA measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .838, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PROMIS: EDA measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .890, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

11. Other Pre Specified Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Baseline Patient Reported Outcomes Measurement Information System (PROMIS): Ability to Participate in Social Roles and Activities Short Form (PROMIS: APRA)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. The PROMIS: APRA is a 4-item questionnaire that measures the perceived ability to perform one's everyday social roles and activities. Scores range 4-20 with higher scores representing fewer limitations (greater abilities).
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: PROMIS: APRA = 5 | 0.57 [0.35 to 0.80] | 0.46 [0.23 to 0.70]
  Baseline to 8 Weeks: PROMIS: APRA = 10 | 0.74 [0.60 to 0.89] | 0.73 [0.58 to 0.88]
  Baseline to 8 Weeks: PROMIS: APRA = 15 | 0.91 [0.69 to 1.13] | 1.00 [0.77 to 1.24]
  Baseline to 20 Weeks: PROMIS: APRA = 5 | 0.33 [0.23 to 0.44] | 0.24 [0.13 to 0.34]
  Baseline to 20 Weeks: PROMIS: APRA = 10 | 0.40 [0.33 to 0.47] | 0.32 [0.25 to 0.40]
  Baseline to 20 Weeks: PROMIS: APRA = 15 | 0.47 [0.36 to 0.58] | 0.41 [0.30 to 0.53]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PROMIS: APRA measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .425, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; PROMIS: APRA measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .733, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

12. Other Pre Specified Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Baseline Five Facet Mindfulness Questionnaire (FFMQ) Abbreviated
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. The FFMQ is a 39-item questionnaire that examines five aspects of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Only the questions related to non-judging of inner experience and non-reactivity were administered (15 items total). The total score on these 15 items was used (range: 15-75). Higher scores represent greater mindfulness.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: FFMQ = 40 | 1.06 [0.85 to 1.26] | 0.97 [0.75 to 1.19]
  Baseline to 8 Weeks: FFMQ = 50 | 0.78 [0.64 to 0.93] | 0.75 [0.60 to 0.90]
  Baseline to 8 Weeks: FFMQ = 60 | 0.51 [0.32 to 0.70] | 0.53 [0.34 to 0.73]
  Baseline to 20 Weeks: FFMQ = 40 | 0.52 [0.42 to 0.62] | 0.41 [0.31 to 0.52]
  Baseline to 20 Weeks: FFMQ = 50 | 0.41 [0.34 to 0.48] | 0.33 [0.25 to 0.40]
  Baseline to 20 Weeks: FFMQ = 60 | 0.30 [0.22 to 0.39] | 0.24 [0.15 to 0.33]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; FFMQ measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .582, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; FFMQ measured at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .666, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

13. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Self-Reported Presence of Psychiatric Illness (Yes or No)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Participants reported whether they have a psychiatric illness.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: Psychiatric Illness | 0.86 [0.59 to 1.13] | 0.68 [0.40 to 0.96]
  Baseline to 8 Weeks: No Psychiatric Illness | 0.75 [0.57 to 0.92] | 0.79 [0.60 to 0.97]
  Baseline to 20 Weeks: Psychiatric Illness | 0.86 [0.86 to 0.86] | 0.68 [0.68 to 0.68]
  Baseline to 20 Weeks: No Psychiatric Illness | 0.37 [0.29 to 0.46] | 0.32 [0.24 to 0.41]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Presence of psychiatric illness at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .355, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Presence of psychiatric illness at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .361, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

14. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Self-Reported Presence of Medical Problems (Yes or No)
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Participants reported whether they have a major medical problem.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: Medical Problems | 0.79 [0.62 to 0.96] | 0.80 [0.61 to 0.98]
  Baseline to 8 Weeks: No Medical Problems | 0.78 [0.50 to 1.06] | 0.67 [0.38 to 0.96]
  Baseline to 20 Weeks: Medical Problems | 0.79 [0.79 to 0.79] | 0.80 [0.80 to 0.80]
  Baseline to 20 Weeks: No Medical Problems | 0.38 [0.25 to 0.52] | 0.37 [0.24 to 0.51]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Presence of medical problems at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .640, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Presence of medical problems at the beginning of the intervention period was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .396, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

15. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Percentage of Sessions Completed
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Percentage of total study sessions completed was calculated.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: 0% | 0.27 [0.03 to 0.51] | 0.64 [0.37 to 0.90]
  Baseline to 8 Weeks: 33% | 0.61 [0.45 to 0.77] | 0.70 [0.52 to 0.87]
  Baseline to 8 Weeks: 100% | 1.28 [1.02 to 1.55] | 0.82 [0.57 to 1.07]
  Baseline to 20 Weeks: 0% | 0.26 [0.14 to 0.37] | 0.26 [0.14 to 0.39]
  Baseline to 20 Weeks: 33% | 0.35 [0.27 to 0.42] | 0.31 [0.22 to 0.39]
  Baseline to 20 Weeks: 100% | 0.53 [0.41 to 0.65] | 0.39 [0.28 to 0.51]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Percentage of sessions completed was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .004, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Percentage of sessions completed was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .291, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

16. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Education
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Participants reported their level of education.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: High School or Less | 0.38 [-0.35 to 1.11] | 0.39 [-0.31 to 1.08]
  Baseline to 8 Weeks: 2 or 4-Year College | 0.84 [0.63 to 1.06] | 0.75 [0.53 to 0.97]
  Baseline to 8 Weeks: > College | 0.73 [0.52 to 0.95] | 0.87 [0.64 to 1.10]
  Baseline to 20 Weeks: High School or Less | 0.40 [0.06 to 0.75] | 0.20 [-0.15 to 0.55]
  Baseline to 20 Weeks: 2 or 4-Year College | 0.44 [0.34 to 0.54] | 0.31 [0.20 to 0.41]
  Baseline to 20 Weeks: > College | 0.37 [0.27 to 0.46] | 0.37 [0.27 to 0.48]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Level of education was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .603, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Level of education was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .333, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

17. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Race
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Participants reported their race.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: White | 0.82 [0.66 to 0.97] | 0.77 [0.61 to 0.94]
  Baseline to 8 Weeks: Non-White | 0.29 [-0.28 to 0.87] | 0.78 [0.20 to 1.35]
  Baseline to 20 Weeks: White | 0.40 [0.33 to 0.47] | 0.34 [0.26 to 0.41]
  Baseline to 20 Weeks: Non-White | 0.41 [0.15 to 0.67] | 0.37 [0.10 to 0.64]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Race was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .224, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = .885, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

18. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Sex
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Participants reported sex assigned at birth.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: Male | 0.49 [0.18 to 0.81] | 0.51 [0.17 to 0.84]
  Baseline to 8 Weeks: Female | 0.85 [0.68 to 1.01] | 0.82 [0.65 to 1.00]
  Baseline to 8 Weeks: Other | 1.85 [-0.22 to 3.91] | 0.18 [-1.58 to 1.94]
  Baseline to 20 Weeks: Male | 0.27 [0.13 to 0.41] | 0.27 [0.12 to 0.42]
  Baseline to 20 Weeks: Female | 0.45 [0.37 to 0.52] | 0.35 [0.26 to 0.43]
  Baseline to 20 Weeks: Other | 1.29 [0.34 to 2.24] | 0.34 [-0.42 to 1.10]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Sex was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .490, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Sex was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .266, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

19. Post Hoc Outcome: Estimated Weekly Change in World Health Organization-5 (WHO-5) Stratified by Ethnicity
Description: The WHO-5 is a 5-item questionnaire that assesses well-being over the prior two weeks. Scores range 0-100 with higher scores reflecting greater well-being. Participants reported their ethnicity.
Time Frame: Baseline to 8 Weeks, Baseline to 20 Weeks
Measure: Mean (95% Confidence Interval); unit: estimated weekly change in WHO-5 score
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
Number analyzed (Participants) | 2220 | 2192
estimated weekly change in WHO-5 score
  Baseline to 8 Weeks: Hispanic | 0.92 [0.12 to 1.71] | 0.88 [0.13 to 1.63]
  Baseline to 8 Weeks: Non-Hispanic | 0.76 [0.61 to 0.91] | 0.77 [0.61 to 0.93]
  Baseline to 8 Weeks: Other | 0.67 [-3.14 to 4.48] | 0.68 [-3.12 to 4.49]
  Baseline to 20 Weeks: Hispanic | 0.56 [0.17 to 0.95] | 0.23 [-0.13 to 0.58]
  Baseline to 20 Weeks: Non-Hispanic | 0.40 [0.33 to 0.47] | 0.34 [0.27 to 0.41]
  Baseline to 20 Weeks: Other | 0.74 [-2.60 to 4.08] | 0.68 [-2.66 to 4.02]
Statistical Analysis 1: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Ethnicity was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 8; Test type: Superiority; p = .928, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction
Statistical Analysis 2: Comparison: Mindfulness-Based Cognitive Therapy vs Brief Mindfulness; Ethnicity was analyzed as a moderator of the relationship between treatment and weekly WHO-5 scores. We added a main effect for the moderator, as well as treatment by time, moderator by time, and treatment by moderator by time interactions to the linear mixed model and used a likelihood ratio test to compare this interaction model to one without the three-way interaction. These analyses were completed over Baseline to Week 20; Test type: Superiority; p = .307, Mixed Models Analysis — Reported p-value is for estimated weekly change in WHO-5 score by treatment by moderator interaction

ADVERSE EVENTS:
Time Frame: 20 weeks.
Description: Data on adverse events (AEs) were collected with a 3-item questionnaire at all study sessions after study randomization. Participants provided a written description of the event, and three study staff sorted these into appropriate organ systems: two coded responses independently and the third resolved discrepancies. Participants reported the event severity, based on a plain-English definition of a serious adverse event (SAE). No AEs/SAEs were reported by participants to be study-related.
Arm/Group | Mindfulness-Based Cognitive Therapy | Brief Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/2220 | 0/2192
Serious Adverse Events (participants affected / at risk) | 30/2220 | 31/2192
Other Adverse Events (participants affected / at risk) | 33/2220 | 41/2192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Cognitive Therapy (N=2220) | Brief Mindfulness (N=2192)
Cardiac Issue (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal Issue (Gastrointestinal disorders) | 3 (3) | 6 (6)
Undefined Health Issue (General disorders) | 2 (2) | 4 (4)
Immune System Issue (Immune system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal or Connective Tissue Issue (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6)
Nervous System Issue (Nervous system disorders) | 3 (3) | 0 (0)
Psychiatric Issue (Psychiatric disorders) | 1 (1) | 2 (2)
Renal Issue (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory Issue/Flu (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Negative Life Event (Social circumstances) | 10 (10) | 10 (11)
Surgical or Medical Procedure (Surgical and medical procedures) | 3 (3) | 1 (1)
Blood/Lymphatic Issue (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Cognitive Therapy (N=2220) | Brief Mindfulness (N=2192)
Cardiac Issue (Cardiac disorders) | 1 (1) | 1 (1)
Endocrine Issue (Endocrine disorders) | 0 (0) | 1 (1)
Gastrointestinal Issue (Gastrointestinal disorders) | 4 (4) | 10 (14)
Undefined Health Issue (General disorders) | 5 (6) | 9 (10)
Injury or Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Musculoskeletal or Connective Tissue Issue (Musculoskeletal and connective tissue disorders) | 9 (10) | 9 (9)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Nervous System Issue (Nervous system disorders) | 5 (6) | 1 (1)
Medication Side-Effect (Product Issues) | 1 (1) | 1 (1)
Psychiatric Issue (Psychiatric disorders) | 2 (2) | 1 (1)
Renal Issue (Renal and urinary disorders) | 0 (0) | 3 (3)
Respiratory Issue/Flu (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin Condition (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Negative Life Event (Social circumstances) | 1 (1) | 2 (2)
Surgical or Medical Procedure (Surgical and medical procedures) | 1 (1) | 1 (2)
Vascular Issue (Vascular disorders) | 0 (0) | 1 (1)
Blood or Lymphatic Issue (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Vision/Eye Issue (Eye disorders) | 1 (1) | 0 (0)
Immune System Issue (Immune system disorders) | 2 (2) | 0 (0)
Injury or Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Reproductive Issue (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Despite having a wide range of clinical and non-clinical samples represented in this study, the sample generalizability was limited in regards to race and gender. A second limitation was not including support for participants to access the study (e.g., technical support, translated versions into other languages) as well as to engage with the study interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03844321/Prot_SAP_000.pdf